CLINICAL TRIAL: NCT03930888
Title: Nutritional Support and Its Influence on the Reduction of Muscle Strength, Muscle Mass and Self-sufficiency in Patients Undergoing Surgical Treatment of Colorectal Cancer
Brief Title: Nutritional Support in Patients Undergoing Surgical Treatment of Colorectal Cancer
Acronym: NISS
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: CHIR-04-NISS
Record Dates: First submitted 2019-04-09; First posted 2019-04-29 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Colorectal Cancer
Keywords: nutritional support; colorectal cancer; muscle strength; muscle mass; self-sufficiency
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with nutritional support: Evaluation of changes in muscle strength, muscle mass and self-sufficiency (ADL-Activites of Daily Living) over a 5-day time period in patients nutritionally supported by nutritional supplements.
  Interventions: Dietary Supplement: Dietary supplement
- Patients without nutritional support: Evaluation of changes in muscle strength, muscle mass and self-sufficiency (ADL-Activites of Daily Living) over a 5-day time period in patients without special nutritional supplements.
  Interventions: Dietary Supplement: Dietary supplement

INTERVENTIONS:
Dietary Supplement: Dietary supplement — Patients with preoperative nutritional support with special nutritional supplements vs. patients without special nutritional support.

SUMMARY:
According to available data, 30-60% of patients are undernourished at hospital admission. The significance of the perioperative nutrition has already been studied in the 1930s. The outcomes of published studies demonstrated that patients with basic nutrient deficiencies have a higher frequency of postoperative complications and have a significantly longer recovery period.

The main aim of the this prospective clinical trial is to evaluate the loss of muscle mass and strength of the patient, the self-sufficiency and the possibility of returning to normal activities, in relation to pre-operatively served nutritional supplements in patients undergoing elective surgery for colorectal cancer.

DETAILED DESCRIPTION:
Malnutrition is a pathological condition of the body caused by a deficiency of essential nutrients. The main feature is protein deficiency, which is caused by disruption of protein and energy balance and needs in the body. According to available data, 30-60% of patients are undernourished at hospital admission. The significance of the perioperative nutrition has already been studied in the 1930s. The outcomes of published studies demonstrated that patients that patients with basic nutrient deficiencies have a higher frequency of postoperative complications and have a significantly longer recovery period.

In 1992, a randomized clinical trial "Peri-operative nutritional support" showed that 85% of hospitalized seniors have malnutrition. The study demonstrated the need for nutritional training to prevent complications and clearly showed a relationship between malnutrition and reconvalescence length and mortality rate. In 2004, another large randomized trial ("Randomized clinical trial of the effects of preoperative and post operative oral nutritional supplements on clinical course and cost of care") confirmed the relationship between malnutrition and the incidence of all perioperative complications. Several other studies, which have been realized within the last decade, confirmed the positive effect of good nutritional condition on postoperative morbidity and mortality.

To the best of the investigator's knowledge, all clinical trials dealing with the issue of preoperative nutrition (published up to now) were primarily focused on the research of the relationship between malnutrition and the frequency of postoperative complications.

The main aim of the this prospective clinical trial is to evaluate the loss of muscle mass and strength of the patient, the self-sufficiency and the possibility of returning to normal activities, in relation to pre-operatively served nutritional supplements in patients undergoing elective surgery for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* resection of colon or rectum due to colorectal cancer

Exclusion Criteria:

* generalization of the disease
* intestinal co-morbidity
* duplicate malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing resection of colon or rectum due to colorectal cancer.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in muscle strength | 6 days
  Muscle strength will be measured in kilograms and changes over a 5-6 day time period in patients nutritionally supported by nutritional supplements and patients without special nutritional supplements will be analysed.
Comparison of muscle mass | 6 days
  Muscle mass will be measured in % of whole body weight and changes over a 5-6 day time period in patients nutritionally supported by nutritional supplements and patients without special nutritional supplements will be analysed.
Self sufficiency | 6 days
  Self sufficiency will be analysed by Barthel Index for Activities of Daily Living, and changes over a 5-6 day time period in patients nutritionally supported by nutritional supplements and patients without special nutritional supplements will be analysed.
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing ADL and mobility. The amount of time and physical assistance required to perform each item are used in determining the assigned value of each item. The total score is 0-100. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital.
Progression of the muscle strength | 6 days
  Muscle strength will be measured in kilograms. The comparison of muscle strength and its progression within 5-6 days between patients with malnutrition and patients in a nutritionally optimal status at hospital admission will be analysed, in relation to patients nutritionally supported by nutritional supplements and patients without special nutritional supplements.
Progression of the muscle mass | 6 days
  Muscle mass will be measured in % of whole body weight. The comparison of muscle mass and its progression within 5-6 days between patients with malnutrition and patients in a nutritionally optimal status at hospital admission will be analysed, in relation to patients nutritionally supported by nutritional supplements and patients without special nutritional supplements.
Progression of the self sufficiency | 6 days
  Self sufficiency will be analysed by Barthel Index for Activities of Daily Living. The comparison of self sufficiency and its progression within 5-6 days between patients with malnutrition and patients in a nutritionally optimal status at hospital admission will be analysed, in relation to patients nutritionally supported by nutritional supplements and patients without special nutritional supplements.
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing ADL and mobility. The amount of time and physical assistance required to perform each item are used in determining the assigned value of each item. The total score is 0-100. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital.

SECONDARY OUTCOMES:
Nutrition status | 1 days
  Nutrition status will be measured by value of concentrations of albumin and prealbumin (transthyretin) in g/l at day of hospital admission. The comparison of the nutrition status in patients with/without preoperative nutritional supplements will be analysed.
Effect of tumor localization | 6 days
  The evaluation whether tumor localization (colon caecum, ascendens, flexura hepatica, colon transversum, flexura lienalis, colon descendens, sigmoideum rectum, anus) affects the pre-operative nutrition status of the patient's (will be measured by value of concentrations of albumin and prealbumin (transthyretin) in g/l at day of hospital admission) and subsequently post-operative progression.

CONTACTS AND LOCATIONS:
Overall Officials: Milan Tesař, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region,, Czechia

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Manasek V, Bezdek K, Foltys A, Klos K, Smitka J, Smehlik D. The Impact of High Protein Nutritional Support on Clinical Outcomes and Treatment Costs of Patients with Colorectal Cancer. Klin Onkol. 2016 Fall;29(5):351-357. PMID 27739314
- [Background] Gillis C, Buhler K, Bresee L, Carli F, Gramlich L, Culos-Reed N, Sajobi TT, Fenton TR. Effects of Nutritional Prehabilitation, With and Without Exercise, on Outcomes of Patients Who Undergo Colorectal Surgery: A Systematic Review and Meta-analysis. Gastroenterology. 2018 Aug;155(2):391-410.e4. doi: 10.1053/j.gastro.2018.05.012. Epub 2018 May 8. PMID 29750973
- [Background] Bruns ERJ, Argillander TE, Van Den Heuvel B, Buskens CJ, Van Duijvendijk P, Winkels RM, Kalf A, Van Der Zaag ES, Wassenaar EB, Bemelman WA, Van Munster BC. Oral Nutrition as a Form of Pre-Operative Enhancement in Patients Undergoing Surgery for Colorectal Cancer: A Systematic Review. Surg Infect (Larchmt). 2018 Jan;19(1):1-10. doi: 10.1089/sur.2017.143. Epub 2017 Oct 19. PMID 29049000
- [Background] Tanaka T, Sato T, Yamashita K, Hosoda K, Nakamura T, Watanabe M. Effect of Preoperative Nutritional Status on Surgical Site Infection in Colorectal Cancer Resection. Dig Surg. 2017;34(1):68-77. doi: 10.1159/000448123. Epub 2016 Jul 28. PMID 27463391
- [Background] Yamano T, Yoshimura M, Kobayashi M, Beppu N, Hamanaka M, Babaya A, Tsukamoto K, Noda M, Matsubara N, Tomita N. Malnutrition in rectal cancer patients receiving preoperative chemoradiotherapy is common and associated with treatment tolerability and anastomotic leakage. Int J Colorectal Dis. 2016 Apr;31(4):877-84. doi: 10.1007/s00384-016-2507-8. Epub 2016 Feb 18. PMID 26888783
- [Derived] Tesar M, Kozusnikova V, Martinek L, Durdik S, Ihnat P. Preoperative nutritional support for patients undergoing elective colorectal cancer surgery - does it really work? Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2023 Jun;167(2):145-151. doi: 10.5507/bp.2022.009. Epub 2022 Mar 1. PMID 35258042